CLINICAL TRIAL: NCT03864562
Title: Gastric Emptying in Non-diabetic Individuals With Black African/Caribbean Heritage - Implications for the Pathogenesis of Type 2 Diabetes
Brief Title: Gastric Emptying - Implications for the Pathogenesis of Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: University of Adelaide (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Other Study IDs: 226-1901
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: gastric emptying; oral glucose tolerance test; Ethnicity; Diabetes risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Black African or Caribbean: Healthy individuals of black African or Caribbean descent
- White European: Healthy individuals of white European descent

SUMMARY:
People of black African and Caribbean descent have a greater risk of developing type 2 diabetes than white Europeans. The aim of this study is to increase our knowledge of how the condition may arise, and what underlies this increased risk. Following a successful screening visit to confirm eligibility for the study, we will be investigating how quickly a glucose drink empties out of the stomach in 30 white Europeans and 30 people of black African or Caribbean descent. In addition, we will study the impact that gastric emptying rate has on blood glucose and satiety hormones released normally by the gut in response to eating. Blood and breath samples will be collected before and during an oral glucose tolerance test.

DETAILED DESCRIPTION:
Background It is recognized that there are differences between ethnic groups in the risk of developing type 2 diabetes (T2D), but the underlying pathophysiology remains poorly defined. For example, whilst insulin resistance, exacerbated by obesity, is common in Caucasian, Hispanic and South Asian populations, impairment in insulin secretion appears to be the primary defect in the pathogenesis of T2D in East Asians. Within the United Kingdom (UK), diabetes and its complications disproportionately affect ethnic minority groups, particularly those of black African-Caribbean (AfC) descent. Studies indicate that the rate of gastric emptying is a major determinant of postprandial glycemia and insulinemia in those with a White European (WE) background in both health and T2D, and although there is evidence that gastric emptying is influenced by ethnicity (which may contribute to the development of T2D), gastric emptying has, to our knowledge, not been evaluated in those of AfC heritage.

Aims The primary objective is to compare the gastric emptying rate in 2 UK ethnic groups. This will be done by conducting a descriptive, cross-sectional pilot study in 60 healthy participants. Secondary objectives are to determine any relationship between glycemia, insulinemia and incretin hormone secretion in these groups.

Experimental protocol Sixty volunteers; 30 of WE and 30 of black AfC heritage will be recruited. Following a successful medical screening visit, participants will be asked to record their dietary intake over 3 days before attending the laboratory for their study visit. On the day before the study visit they will be asked to avoid strenuous exercise, alcohol and caffeine intake and to eat their normal diet. On the study day, participants will arrive at the laboratory in the morning following an overnight fast. A cannula will be inserted into a vein in the top of the hand and the hand placed in a warming box for repeat arterialized-venous blood sampling over the study day. After baseline breath and blood samples have been taken, participants will then be given a drink containing 75g of glucose dissolved in 300ml water (standard oral glucose tolerance test), to which has been added 150mg of 13C labelled acetate, and asked to consume it within 5 minutes. The stable isotope label on the acetate allows us to assess gastric emptying by detecting the appearance of 13CO2 in breath. Blood samples (6ml) will be collected prior to the drink, with further samples being taken every 15min for the first 2hrs, then every 30min for the next hour, with a final sample taken at 4hrs. Blood will be analysed for glucose, insulin, C-peptide, Glucagon-like peptide 1 (GLP-1), glucagon, and Gastric inhibitory polypeptide (GIP). Following the drink, subjects will also be asked to complete satiety and GI symptom questionnaires every half hour throughout the study. At the end of the 4 hours, participants will be asked to complete a series of autonomic function tests, during which we will measure blood pressure and heart rate. These tests are 2mins of rhythmic breathing (5sec inhale: 5sec exhale) and postural change to standing from resting semi-supine. After this time, the cannula will be removed and the study is completed

ELIGIBILITY:
Inclusion Criteria:

* White European or black African / Caribbean heritage
* BMI >18 kg/m2
* Ability to give written informed consent
* English speaking

Exclusion Criteria:

* Any significant medical condition
* Uncontrolled hypertension
* Alcohol consumption >14 units / week
* Random blood Glucose concentration above 7.8mmol/l
* Hemoglobin A1c (HbA1c) >47mmol/mol (>6.4%)
* Use of regular medication, (oral contraceptive pill or antihypertensive medication are acceptable if use has been for >6 months)
* History of Irritable Bowel Syndrome, food intolerances or any gastrointestinal disorders
* Previous bariatric surgery, or gastrointestinal surgery which may affect normal function (e.g. bowel resection)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study cohort will be recruited from the general population of England who live within commuting distance from the study site, and will incorporate those from the counties of Nottinghamshire, Derbyshire and Leicestershire
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Gastric emptying rate | 4 hours
  Time for clearance of half of the glucose drink (measured via a stable isotope breath test and area under the incremental postprandial blood glucose response curve)

SECONDARY OUTCOMES:
Serum Insulin concentration | 4 hours
  Serum Insulin response to the glucose drink, measured by serial blood sampling and later analysis using a radio-immuno assay (RIA)
Whole blood glucose concentration | 4 hours
  Blood glucose response to the glucose drink, measured by serial blood sampling and immediate analysis using the glucose oxidase method
Plasma glucagon concentration | 4 hours
  Plasma glucagon response to the glucose drink, measured by serial blood sampling and later analysis using an RIA
Plasma GLP-1 concentration | 4 hours
  Plasma GLP-1 response to the glucose drink, measured by serial blood sampling and later analysis using an enzyme-linked immunosorbent assay (ELISA)
Plasma GIP concentration | 4 hours
  Plasma GIP response to the glucose drink, measured by serial blood sampling and later analysis using an enzyme-linked immunosorbent assay (ELISA)
Serum C-peptide concentration | 4 hours
  Serum C-peptide response to the glucose drink, measured by serial blood sampling and later analysis using an enzyme-linked immunosorbent assay (ELISA)
Attrition rate | 1 year
  Number of participants completing the protocol as a proportion of those who were recruited to the study
Recruitment rate | 1 year
  Number of people volunteering to take part in the study as a proportion of those expressing initial interest

CONTACTS AND LOCATIONS:
Overall Officials: Michael Horowitz, MD PhD, Study Director — University of Adelaide
Locations (1):
- David Greenfield Human Physiology Unit, University of Nottingham, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kodama K, Tojjar D, Yamada S, Toda K, Patel CJ, Butte AJ. Ethnic differences in the relationship between insulin sensitivity and insulin response: a systematic review and meta-analysis. Diabetes Care. 2013 Jun;36(6):1789-96. doi: 10.2337/dc12-1235. PMID 23704681
- [Background] Horowitz M, Edelbroek MA, Wishart JM, Straathof JW. Relationship between oral glucose tolerance and gastric emptying in normal healthy subjects. Diabetologia. 1993 Sep;36(9):857-62. doi: 10.1007/BF00400362. PMID 8405758
- [Background] Phillips WT. Gastric emptying in ethnic populations: possible relationship to development of diabetes and metabolic syndrome. Ethn Dis. 2006 Summer;16(3):682-92. PMID 16937605